CLINICAL TRIAL: NCT04317820
Title: The Effects of Deep Brain Reorienting (DBR) on Post-traumatic Stress Disorder (PTSD)
Brief Title: Deep Brain Reorienting in Post-traumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ruth Lanius, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8997; 114501 (Other: Western University's Human Research Ethics)
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: PTSD; Post-traumatic Stress Disorder
Keywords: Deep Brain Reorienting; DBR
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the DBR treatment or wait-list conditions.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blinded to which condition the participant was assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBR Condition (Experimental): Involves 8 weekly sessions of DBR treatment.
  Interventions: Behavioral: Deep Brain Reorienting (DBR)
- Wait-list Condition (No Intervention): No intervention for approximately 8 weeks.

INTERVENTIONS:
Behavioral: Deep Brain Reorienting (DBR) — Trauma processing through DBR involves bringing up a traumatic memory and encouraging the client to focus on tensions arising in the muscles of the shoulders, neck, head and face (i.e., those involved in orienting toward a threatening person/event). The rationale is as follows: Physiologically, orienting to a stimulus, whether external or in the mind's eye, comes before any affective response to it. Here, it is hypothesized that there is activity in certain midbrain structures , i.e.,Superior Colliculi (SC) and Periaqueductal Gray (PAG). The deep layers of the SC bring on a brief (orienting) tension in the neck as well as preparing for eye movements, which is later followed by the processing of raw affect in the PAG. In session, if we can attend to this tension - even if we have to backtrack from the emotion that follows - we can establish an anchor in the body that precedes the affect and is hypothesized to protect against emotional overwhelm.
  Arms: DBR Condition

SUMMARY:
This study will evaluate the efficacy of a therapeutic treatment, Deep Brain Reorienting (DBR), for PTSD (Post-traumatic Stress Disorder). Participants will be randomized to either the DBR treatment, or wait-list condition.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of Deep Brain Reorienting (DBR) in reducing PTSD symptoms. DBR was designed by Dr. Frank Corrigan, a Scottish psychiatrist interested in the brain mechanisms underlying effective trauma psychotherapy. For this study, participants will be randomized to either the DBR treatment or wait-list study conditions. Trauma processing through DBR involves bringing up a traumatic memory and encourages the client to focus on tensions arising in the muscles of the shoulders, neck, head and face (i.e., those involved in orienting toward a threatening person/event). It is believed that this approach will allow the participant to process the traumatic memory in an emotionally manageable way, changing how it is represented/accessed in the brain's innate defensive system. Online Stream - Assessments will include clinical interviews (pre/post treatment, and follow-up) using Webex video conferencing, and fMRI (functional magnetic resonance imaging) scans (pre/post treatment). In-Person Stream - Assessment will include clinical interviews (pre/post treatment and follow-up), and fMRI scans (pre/post treatment).

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* age: 18-65
* meets diagnostic criteria for PTSD (as determined by study assessment)
* may benefit from short-term trauma therapy (as determined by study assessment)

Exclusion Criteria:

* Individuals with any implants, conditions, etc. that do not comply with 7-Tesla (7T) fMRI research safety standards (e.g., certain implants, pregnancy)
* history of significant head injury/lengthy loss of consciousness (e.g., a Glasgow Coma Scale Score < 15 at the time of incident assessed retrospectively by participant)
* significant untreated medical illness
* history of neurological disorder
* history of any pervasive developmental disorder
* history of bipolar disorder
* history of psychotic disorder
* alcohol/substance abuse or dependence within the last 3 months
* extensive narcotic use
* current participation in counselling more extensive than supportive therapy (e.g., exposure therapy, Cognitive-Behavioural Therapy would be an exclusion)
* a degree of mental distress that is unlikely to benefit from a short-term therapy (for our participants' well-being, it will be necessary that we believe it possible to safely address the issues/triggers brought up in treatment within the 8 sessions).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
change in PTSD symptoms from baseline as measured by the Clinician Administered PTSD Scale (CAPS) at post-treatment assessment | 8 weeks
  min. CAPS score=0, max=80, with higher scores representing greater PTSD symptoms
change in PTSD symptoms from post-treatment assessment as measured by the Clinician Administered PTSD Scale (CAPS) at follow-up assessment | 3 months
  min. CAPS score=0, max=80, with higher scores representing greater PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Lanius, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corneil BD, Munoz DP, Chapman BB, Admans T, Cushing SL. Neuromuscular consequences of reflexive covert orienting. Nat Neurosci. 2008 Jan;11(1):13-5. doi: 10.1038/nn2023. Epub 2007 Dec 2. PMID 18059264
- [Background] Lanius RA, Rabellino D, Boyd JE, Harricharan S, Frewen PA, McKinnon MC. The innate alarm system in PTSD: conscious and subconscious processing of threat. Curr Opin Psychol. 2017 Apr;14:109-115. doi: 10.1016/j.copsyc.2016.11.006. Epub 2016 Nov 26. PMID 28813307
- [Background] Terpou BA, Densmore M, Thome J, Frewen P, McKinnon MC, Lanius RA. The Innate Alarm System and Subliminal Threat Presentation in Posttraumatic Stress Disorder: Neuroimaging of the Midbrain and Cerebellum. Chronic Stress (Thousand Oaks). 2019 Feb 5;3:2470547018821496. doi: 10.1177/2470547018821496. eCollection 2019 Jan-Dec. PMID 32440590
- [Background] Comoli E, Das Neves Favaro P, Vautrelle N, Leriche M, Overton PG, Redgrave P. Segregated anatomical input to sub-regions of the rodent superior colliculus associated with approach and defense. Front Neuroanat. 2012 Apr 3;6:9. doi: 10.3389/fnana.2012.00009. eCollection 2012. PMID 22514521
- [Derived] Kearney BE, Corrigan FM, Frewen PA, Nevill S, Harricharan S, Andrews K, Jetly R, McKinnon MC, Lanius RA. A randomized controlled trial of Deep Brain Reorienting: a neuroscientifically guided treatment for post-traumatic stress disorder. Eur J Psychotraumatol. 2023;14(2):2240691. doi: 10.1080/20008066.2023.2240691. PMID 37581275